CLINICAL TRIAL: NCT05589194
Title: The Effect of Comfort Theory-Based Nursing Interventions on Urinary Incontinence, Quality of Life, and Comfort Levels in Women with Stress Urinary Incontinence: a Randomized Controlled Study
Brief Title: Comfort Theory-Based Nursing Interventions in Women with Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hilal Gamze Hakbilen, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AkdenizNursing
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-07

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Comfort Theory; Yoga; Nursing
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled single-blind quasi-experimental research design.
Who Masked: Participant
Masking Description: In the randomization process, those who meet the criteria for inclusion in the sample and accept to participate in the study do not know that they will be included in the intervention group or the control group, so it will be single-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): After the first interview with the patients in the intervention group, a phone call will be made for regarding the implementation of nursing interventions based on the Comfort Theory, and they will be informed about the planned dates for the implementation. The implementation phase of nursing interventions based on Comfort Theory will be carried out for 6 weeks at the Communication Laboratory of the Faculty of Nursing of Akdeniz University on the planned dates with the patients. In addition, a handbook will be given to the patients at the beginning of the practice, and the Home Yoga Diary in the handbook will be expected to be filled in daily by the patients during the research. Immediately after the implementation of the nursing interventions based on Comfort Theory (week 6), patients will be asked to fill in ISI, IQO-L, and the Urinary Incontinence and Frequency Comfort Scale. During this whole process, patients will continue their planned routine care and treatment.
  Interventions: Behavioral: Nursing Practices Based on Kolcaba's Comfort Theory
- Control Group (No Intervention): After the first interview with the patients in the control group, the routine care and treatment practices planned by the polyclinic physician and nurse will continue. No additional intervention is planned for the patients in this group. A new interview will be planned with the patients in the control group 6 weeks after the first interview, and they will be asked to fill in the ISI, IQO-L, and the Urinary Incontinence and Frequency Comfort Scale.

INTERVENTIONS:
Behavioral: Nursing Practices Based on Kolcaba's Comfort Theory — Nursing interventions planned to be carried out within the scope of the research will be based on Comfort Theory. Nursing interventions will be planned according to the needs in the physical comfort (diet practice, providing effective and correct pelvic floor muscle contraction, repetitive and regular yoga practice training), psychospiritual comfort (appreciation and encouragement, self-confidence, expressing the feeling of embarrassment, expressing fear, confidence, repetitive and regular practice of yoga practice, meditation), sociocultural comfort (to be informed, to develop effective interpersonal communication, to interact with other women with SUI) and environmental comfort (Informing about making the necessary arrangements to prevent possible situations such as sleep disruption and falling, bad smell, etc. and performing nursing practices by respecting privacy). The yoga practice will carry out with the participation of 60-minute group yoga classes twice a week for 6 weeks.
  Arms: Intervention Group

SUMMARY:
Urinary incontinence (UI) is a symptom that develops due to damage to the bladder, sphincter mechanism or pelvic floor muscles, defined as unconscious urinary incontinence, which is a common health problem among adult women. Urinary incontinence can be classified as urge incontinence (UUI), stress incontinence (SUI) or mixed incontinence (MUI). Considering the prevalence values of UI subtypes that change with age, it was found that SUI was the highest (32%) in the 40-59 age group.

Although UI is not life-threatening, it imposes significant limitations on women's activities of daily living and sexual and interpersonal relationships. Emotional problems such as embarrassment, depression, sadness and low body image associated with UI have a negative impact on quality of life. Pharmacological, surgical and behavioral treatment methods can be applied in the treatment of UI, which causes significant negative effects on quality of life. However, there are various limitations in the implementation of these methods. This situation has revealed the necessity of developing new methods in the treatment of UI. One of the behavioral treatment methods that can provide therapeutic benefits for urinary incontinence is yoga. Recently, yoga has become a new option for strengthening pelvic floor muscles and treating symptoms related to pelvic floor dysfunctions. Yoga can be practiced by women without constant supervision by healthcare providers, thus providing an accessible and cost-effective self-management strategy for large numbers of women in the community.

Nurses have important roles and responsibilities in the diagnosis, treatment and care process of UI. Nurses need to plan and implement a care that will increase the quality of life and provide comfort for patients with UI. The word comfort, which we often use in our daily life, expresses a basic human need. The taxonomic structure of the Comfort Theory, which was formed on the basis of the concept of comfort, which is a nursing function, attempt and at the same time, the intended result of most nursing interventions, consisting of three levels and four dimensions, was revealed by Kolcaba in 1988. Kolcaba emphasized that comfort care is a process as an attempt to achieve comfort, and that increasing comfort level is a product.

In the literature, no randomized controlled study was found in which nursing interventions based on Comfort Theory were applied to female patients with a diagnosis of SUI. In this study, it is aimed to evaluate the effect of nursing interventions based on Comfort Theory applied to female patients with a diagnosis of SUI on UI, quality of life and comfort level.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is seen as a common health problem among adult women. UI, defined as unconscious urinary incontinence, is not a disease, but a symptom that develops due to damage to the bladder, sphincter mechanism, or pelvic floor muscles. Different rates are expressed regarding the incidence of UI in the world. When population studies conducted in many countries are evaluated, it has been determined that the incidence of UI varies between 5% and 70%. Population-based studies have reported that UI is more common in women than men, and approximately 10% of all adult women experience UI.

Urinary incontinence can be classified as urge incontinence (UII) (involuntary leakage accompanied by urgency), stress incontinence (SUI) (involuntary leakage upon exertion or sneezing or coughing), or mixed incontinence (MUI) (involuntary leakage associated with urgency and effort, sneezing or coughing). In a prevalence study, the prevalence of any type of UI among women was found to be 53%; according to UI subtypes, 16% of women had MUI, 26% had SUI and 10% had UUI. Although many adult women experience SUI today, they see this as a natural consequence of birth and aging and do not think that it is a serious health problem. As a result of this situation, women do not attempt to apply for health services for UI. However, although UI is not life-threatening, it imposes significant limitations on women's activities of daily living and sexual and interpersonal relationships. Emotional problems such as embarrassment, depression, sadness, and low body image that UI brings with it cause a negative effect on quality of life.

Pharmacological, surgical, and behavioral treatment methods can be applied in the treatment of UI, which causes significant negative effects on quality of life. One of the behavioral treatment methods that can provide therapeutic benefits for urinary incontinence is yoga. Yoga is an ancient medical practice used to maintain bodily health and heal many types of diseases. Recently, yoga has become a new option to strengthen the pelvic floor muscles and treat symptoms related to pelvic floor dysfunctions. When the literature is examined, the results of studies showing that yoga practice is very effective in the treatment of UI have been found. Unlike most UI treatments, yoga can be practiced by women without constant supervision from healthcare providers, thus offering an accessible and cost-effective self-management strategy for large numbers of women in the community.

Nurses have important roles and responsibilities in the diagnosis, treatment, and care process of UI. Nurses need to plan and implement a care that will increase the quality of life and provide comfort for patients with UI. The word comfort, which we often use in our daily life, expresses a basic human need. Comfort is a nursing function, initiative, and also the intended outcome of most nursing interventions in the field of nursing. Kolcaba created the taxonomic structure of Comfort Theory, consisting of three levels and four dimensions, in 1988. The 3 levels within the scope of the theory were created depending on the intensity of meeting the individual comfort needs of the patients. In other words, the level of meeting the patients' needs for comfort created 3 levels of the Comfort Theory. These levels are respectively; relief, relief, and superiority. Kolcaba handled Comfort Theory in 4 dimensions taxonomically. These dimensions are based on a holistic philosophy, that is, a holistic perspective, and are named physical comfort, psychospiritual comfort, sociocultural comfort, and environmental comfort. When the taxonomic structure of Comfort Theory is evaluated, it is seen that all its components are interconnected. For example; physical comfort is related to bodily perceptions. When the individual's needs for physical responses to various stimuli are met, the individual will get rid of the distress of these responses and reach the desired comfort level. Kolcaba emphasized that comfort care is a process as an attempt to achieve comfort, and that increasing comfort level is a product.

In the literature, no randomized controlled study was found in which nursing interventions based on Comfort Theory were applied to female patients with SUI. In this study, it is aimed to evaluate the effect of nursing interventions based on Comfort Theory applied to female patients with SUI on UI, quality of life, and comfort level. In addition, it is thought that the results obtained from this study will increase awareness of practices such as yoga, meditation, and breathing exercises as an effective, applicable, and easily adaptable behavioral treatment method in female patients with a diagnosis of SUI.

AIM OF THE STUDY The aim of this study; To examine the effects of nursing interventions based on Comfort Theory applied to female patients with SUI on UI, quality of life and comfort levels.

HYPOTHESES OF THE STUDY

1. H1: Nursing interventions based on Comfort Theory have an effect on the UI level of female patients with SUI.
2. H1: Nursing interventions based on Comfort Theory have an effect on the quality of life of female patients with SUI.
3. H1: Nursing interventions based on Comfort Theory have an effect on the comfort level of female patients with SUI.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* Diagnosed with SUI
* Continuing to experience UI complaints for at least 3 months
* Who agreed to participate in the research

Exclusion Criteria:

* Diagnosed with pelvic organ prolapse
* Experienced urinary tract infection or hematuria more than 3 times in the last 1 year
* Having major neurological health problems
* Pelvic cancer patient
* Having chronic pelvic pain
* BMI>35 kg/m2
* Having a history of urinary system surgery
* Having yoga experience in the last 1 year
* Actively doing pelvic floor exercises
* Have given birth in the last 6 months
* Pregnancy
* Having limited movement
* Alcohol/drug addiction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will be limited to female patients with a diagnosis of SUI.
Enrollment: 40 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Incontinence Severity Index (ISI) | 6 week
  Incontinence Severity Index (ISI) will be used to determine the UI severity of the participants. The ISI is a short scale developed by Sandvik et al., which is easily applied to individuals with urinary incontinence. The ISI is an assessment tool consisting of two questions that evaluate the frequency and amount of incontinence. The result regarding the severity of incontinence is calculated by multiplying the scores obtained from the questions. The results obtained are "Mild" (1 and 2 points), "Moderate" (3, 4 and 6 points), "Severe" (8 and 9 points) and "Very Severe" (12 points) are divided into four groups.

SECONDARY OUTCOMES:
Urinary Incontinence Quality of Life Scale (IQO-L) | 6 week
  The Urinary Incontinence Quality of Life Scale (IQO-L) was developed by Wagner et al. to determine the quality of life of patients with UI. The IQO-L was later re-evaluated by Patrick et al. in 1999. In the process of creating the European versions of the scale, 6 questions were removed with the evaluation of psychometric measurements, and the number of questions was reduced to 22. In the IQO-L, all items are evaluated on a 5-point Likert-type scale (1 = a lot, 2 = a lot, 3 = moderately, 4 = a little, 5 = not at all). The total score calculated on the scale is converted to a scale value from 0 to 100 for better understanding. The IQO-L limiting behaviors (1st,2nd,3rd,4th,10th,11th,13th,20th items), psychological influence (5th,6th,7th,9th,15th. ,16.,17.,21.,22. items) and limiting social life (8.,12.,14.,18.,19). High scores indicate that the quality of life is better than low scores.

OTHER OUTCOMES:
Urinary Incontinence and Frequency Comfort Scale | 6 week
  Urinary Incontinence and Frequency Comfort Scale was developed by Dowd et al. using Kolcaba's General Comfort Scale to evaluate the comfort of individuals with UI and urination problems. The scale includes the comfort of an individual with urinary incontinence in four dimensions: physical, psychospiritual, sociocultural and environmental; It contains 28 expressions that evaluate at three levels as relief, relief, and superiority. Each statement in the scale has a Likert-type rating ranging from 1 to 6 from "Strongly Disagree" to "Strongly Agree". 16 of the expressions are positive (1, 2, 4, 9, 11, 12, 13, 15, 16, 17, 23, 24, 25, 26, 27, 28), 12 negative (3, 5, 6, 7, 8, 10, 14, 18, 19, 20, 21, 22); negative statements are reversed in scoring. The highest total score that can be obtained from the scale is 168, and the lowest score is 28. A low score indicates bad comfort, and a high score indicates good comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Aoki Y, Brown HW, Brubaker L, Cornu JN, Daly JO, Cartwright R. Urinary incontinence in women. Nat Rev Dis Primers. 2017 Jul 6;3:17042. doi: 10.1038/nrdp.2017.42. PMID 28681849
- [Background] Charalambous S, Trantafylidis A. Impact of urinary incontinence on quality of life. Pelviperineology. 2009; 28: 51-53.
- [Background] Hagglund D, Walker-Engstrom ML, Larsson G, Leppert J. Reasons why women with long-term urinary incontinence do not seek professional help: a cross-sectional population-based cohort study. Int Urogynecol J Pelvic Floor Dysfunct. 2003 Nov;14(5):296-304; discussion 304. doi: 10.1007/s00192-003-1077-9. Epub 2003 Aug 29. PMID 14618304
- [Background] Huang AJ, Chesney M, Lisha N, Vittinghoff E, Schembri M, Pawlowsky S, Hsu A, Subak L. A group-based yoga program for urinary incontinence in ambulatory women: feasibility, tolerability, and change in incontinence frequency over 3 months in a single-center randomized trial. Am J Obstet Gynecol. 2019 Jan;220(1):87.e1-87.e13. doi: 10.1016/j.ajog.2018.10.031. Epub 2018 Oct 26. PMID 30595143
- [Background] Huang AJ, Jenny HE, Chesney MA, Schembri M, Subak LL. A group-based yoga therapy intervention for urinary incontinence in women: a pilot randomized trial. Female Pelvic Med Reconstr Surg. 2014 May-Jun;20(3):147-54. doi: 10.1097/SPV.0000000000000072. PMID 24763156
- [Background] Irwin DE, Kopp ZS, Agatep B, Milsom I, Abrams P. Worldwide prevalence estimates of lower urinary tract symptoms, overactive bladder, urinary incontinence and bladder outlet obstruction. BJU Int. 2011 Oct;108(7):1132-8. doi: 10.1111/j.1464-410X.2010.09993.x. Epub 2011 Jan 13. PMID 21231991
- [Background] Kim GS, Kim EG, Shin KY, Choo HJ, Kim MJ. Combined pelvic muscle exercise and yoga program for urinary incontinence in middle-aged women. Jpn J Nurs Sci. 2015 Oct;12(4):330-9. doi: 10.1111/jjns.12072. Epub 2015 Feb 23. PMID 25705816
- [Background] Kim HS. A study on self-esteem, depression, anxiety, and discomfort of daily life due to urinary incontinence in women. Journal of Korean Academy of Psychiatric and Mental Health Nursing. 2001; 10: 98-106.
- [Background] Kolcaba K, DiMarco MA. Comfort Theory and its application to pediatric nursing. Pediatr Nurs. 2005 May-Jun;31(3):187-94. PMID 16060582
- [Background] Kolcaba K. Comfort Theory and Practice: A Vision for Holistic Health Care and Research. New York: Springer Publishing. 2003: 15-49.
- [Background] Kolcaba KY. A taxonomic structure for the concept comfort. Image J Nurs Sch. 1991 Winter;23(4):237-40. doi: 10.1111/j.1547-5069.1991.tb00678.x. PMID 1937522
- [Background] Kolcaba KY. Comfort as process and product, merged in holistic nursing art. J Holist Nurs. 1995 Jun;13(2):117-31. doi: 10.1177/089801019501300203. PMID 7745238
- [Background] Kwon BE, Kim GY, Son YJ, Roh YS, You MA. Quality of life of women with urinary incontinence: a systematic literature review. Int Neurourol J. 2010 Oct;14(3):133-8. doi: 10.5213/inj.2010.14.3.133. Epub 2010 Oct 31. PMID 21179330
- [Background] Lee UJ, Feinstein L, Ward JB, Kirkali Z, Martinez-Miller EE, Matlaga BR, Kobashi KC. Prevalence of Urinary Incontinence among a Nationally Representative Sample of Women, 2005-2016: Findings from the Urologic Diseases in America Project. J Urol. 2021 Jun;205(6):1718-1724. doi: 10.1097/JU.0000000000001634. Epub 2021 Feb 19. PMID 33605795
- [Background] Mills C, Evans A, Rogers T. Is yoga an effective treatment of urinary incontinence in women?. Evidence-Based Practice. 2021; 24(4): 41-42.
- [Background] Milsom I, Gyhagen M. The prevalence of urinary incontinence. Climacteric. 2019 Jun;22(3):217-222. doi: 10.1080/13697137.2018.1543263. Epub 2018 Dec 21. PMID 30572737
- [Background] Milsom I, Altman D, Cartwright R, et al. Epidemiology of urinary incontinence (UI) and other lower urinary tract symptoms (LUTS), pelvic organ prolapse (POP) and anal (AI) incontinence. In: Abrams 22. P, Cardozo L, Wagg A, Wein A, eds. Incontinence. 6th ed. Paris: Health Publications Ltd; 2016:17-24.
- [Background] Nayak G, Kamath A, Kumar PN, Rao A. Effect of yoga therapy on physical and psychological quality of life of perimenopausal women in selected coastal areas of Karnataka, India. J Midlife Health. 2014 Oct;5(4):180-5. doi: 10.4103/0976-7800.145161. PMID 25540568
- [Background] Ozcan M, Kapucu S. Nursing approach in elderly patients with urinary ıncontinence. Journal of Hacettepe University Faculty of Nursing. 2014; 101-109.
- [Background] Parker ME, Smith MC. Nursing Theories And Nursing Practice. Philadelphia: Davis Company. 2010: 389-401.
- [Background] Rathore M, Agrawal S, Nayak PK, Sinha M, Sharma DK, Mitra S. Exploring the significance of
- [Background] Sweta KM, Godbole A, Awasthi HH, Pandey U. Effect of Mula Bandha Yoga in Mild Grade Pelvic Organ Prolapse: A Randomized Controlled Trial. Int J Yoga. 2018 May-Aug;11(2):116-121. doi: 10.4103/ijoy.IJOY_32_17. PMID 29755220
- [Background] Tenfelde S, Tell D, Garfield L, Mathews H, Janusek L. Yoga for Women With Urgency Urinary Incontinence: A Pilot Study. Female Pelvic Med Reconstr Surg. 2021 Jan 1;27(1):57-62. doi: 10.1097/SPV.0000000000000723. PMID 30964762
- [Background] Terzi B, Kaya N. Comfort Theory and analysis. Journal of Anatolia Nursing and Health Sciences. 2017; 20(1): 67-74.
- [Background] Tunuguntla R, Tunuguntla HSGR, Kathuria H, Verma S. Effectiveness of App-Based Yoga of Immortals (YOI) Intervention for Insomnia in Asian Population during Pandemic Restrictions. Int J Environ Res Public Health. 2021 May 26;18(11):5706. doi: 10.3390/ijerph18115706. PMID 34073407
- [Background] Vinchurkar SA, Arankalle DV. Integrating yoga therapy in the management of urinary incontinence: a case report. J Evid Based Complementary Altern Med. 2015 Apr;20(2):154-6. doi: 10.1177/2156587214563311. Epub 2014 Dec 24. PMID 25539839
- [Background] Sandvik H, Hunskaar S, Seim A, Hermstad R, Vanvik A, Bratt H. Validation of a severity index in female urinary incontinence and its implementation in an epidemiological survey. J Epidemiol Community Health. 1993 Dec;47(6):497-9. doi: 10.1136/jech.47.6.497. PMID 8120507
- [Background] Hazar UH, Şirin A. Validity and reliability study of incontinence severity index. Journal Of Adnan Menderes University Medical Faculty. 2008; 9(3): 5-8.
- [Background] Wagner TH, Patrick DL, Bavendam TG, Martin ML, Buesching DP. Quality of life of persons with urinary incontinence: development of a new measure. Urology. 1996 Jan;47(1):67-71; discussion 71-2. doi: 10.1016/s0090-4295(99)80384-7. PMID 8560665
- [Background] Patrick DL, Martin ML, Bushnell DM, Yalcin I, Wagner TH, Buesching DP. Quality of life of women with urinary incontinence: further development of the incontinence quality of life instrument (I-QOL). Urology. 1999 Jan;53(1):71-6. doi: 10.1016/s0090-4295(98)00454-3. PMID 9886591
- [Background] Ozerdoğan N, Kızılkaya NB. The prevalence and risk factors of urinary incontinence and its influence on the quality of life in 20 years or older of women in Eskişehir, Afyon, Kütahya, Bilecik cities. Florence Nightingale Journal of Nursing 2003;51:37-50.
- [Background] Dowd T, Kolcaba K, Steiner R. Using cognitive strategies to enhance bladder control and comfort. Holist Nurs Pract. 2000 Jan;14(2):91-103. doi: 10.1097/00004650-200001000-00013. PMID 12119974
- [Background] Zengin N. Effects of nursing education and behavioral therapy on comfort, pelvic muscle exercise self-efficacy and quality of life among women with urinary incontinence. Marmara University Institute of Health Sciences, PhD Thesis, 2008, Istanbul.